CLINICAL TRIAL: NCT04007796
Title: Improving Sleep and Functioning in Veterans With Posttraumatic Stress Disorder
Brief Title: Apnea and Insomnia Relief Study
Acronym: AIR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D2952-W
Record Dates: First submitted 2019-07-02; First posted 2019-07-05 (Actual); Results first posted 2025-12-08 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: Sleep Apnea Syndromes; Insomnia Disorder; Stress Disorders, Post-Traumatic
Keywords: Sleep Apnea Syndromes; Sleep Apnea, Central; Sleep Apnea, Obstructive; Sleep Initiation and Maintenance Disorders; Insomnia; Insomnia Disorder; Stress Disorders, Post-Traumatic; PTSD; Veterans
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Initiation and Maintenance Disorders; Stress Disorders, Post-Traumatic; Sleep Apnea, Central; Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with participants assigned to one of two treatment groups in parallel for the duration of the study
Who Masked: Outcomes Assessor
Masking Description: The clinical interviewer conducting outcome-related interviews will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Apnea and Insomnia Relief (AIR) (Experimental): This treatment will be offered over six sessions. All appointments will be conducted via telehealth and will last 60 minutes. The main components of the AIR protocol are (a) psychoeducation, (b) motivational interviewing, (c) PAP adherence strategies, and (d) cognitive behavioral therapy for insomnia.
  Interventions: Behavioral: Apnea and Insomnia Relief (AIR)
- Sleep Education (SE) (Active Comparator): This treatment will be offered over six sessions. All appointments will be conducted via telehealth and will last 60 minutes. Topics covered include the sleep cycle, sleep across the lifespan, sleep and the mind, evening activities and the sleep environment, and daytime activities and sleep.
  Interventions: Behavioral: Sleep Education (SE)

INTERVENTIONS:
Behavioral: Apnea and Insomnia Relief (AIR) — This treatment will be offered over six sessions. All appointments will be conducted via telehealth and will last 60 minutes. The main components of the AIR protocol are (a) psychoeducation, (b) motivational interviewing, (c) PAP adherence strategies, and (d) cognitive behavioral therapy for insomnia.
  Arms: Apnea and Insomnia Relief (AIR)
Behavioral: Sleep Education (SE) — This treatment will be offered over six sessions. All appointments will be conducted via telehealth and will last 60 minutes. Topics covered include the sleep cycle, sleep across the lifespan, sleep and the mind, evening activities and the sleep environment, and daytime activities and sleep.
  Arms: Sleep Education (SE)

SUMMARY:
The purpose of this study is to determine whether a behavioral sleep treatment improves functioning and sleep in Veterans with posttraumatic stress disorder (PTSD).

DETAILED DESCRIPTION:
This study is a randomized controlled trial of a behavioral sleep treatment to improve functioning and sleep in Veterans with PTSD, sleep apnea, and insomnia. The treatment is delivered via telehealth (video to home). The primary outcome for this study is quality of life. Other outcomes include sleep-related functioning, PTSD symptom severity, insomnia symptom severity, and CPAP adherence. Participants will also provide treatment feedback to aid in assessment of treatment feasibility and acceptability.

ELIGIBILITY:
Inclusion Criteria:

* Veterans diagnosed with sleep apnea with Apnea Hypopnea Index of at least 5 via sleep study and recommended for PAP therapy
* Meet DSM-5 Criteria for Posttraumatic Stress Disorder or subthreshold Posttraumatic Stress Disorder
* Meet DSM-5 Criteria for Insomnia Disorder
* Willing to attend all treatment and assessment appointments
* English literacy and cognition sufficient to participate in treatment and assessment

Exclusion Criteria:

* Psychosis or manic episode in last 5 years
* Moderate or severe substance use disorder in past 6 months
* Started or ended psychotherapy for a sleep disorder or mental health diagnosis within the last 1 month or plans to discontinue this treatment during the trial
* Started or ended an antidepressant, anxiolytic, or sleep medication with the last 1 month or plans to discontinue this treatment during the trial
* Prominent suicidal or homicidal ideation requiring alternative treatment for patient safety
* Untreated sleep disorders that may interfere with successful treatment (up to discretion of Principal Investigator)
* Having travel of personal plans that would disrupt regular treatment engagement (up to discretion of Principal Investigator)
* Working night shifts or rotating shifts that include night shifts
* Lack of stable housing
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-02-27 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2025-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lizabeth A Goldstein, PhD, Principal Investigator — San Francisco VA Medical Center, San Francisco, CA
Locations (1):
- San Francisco VA Medical Center, San Francisco, CA, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Apnea and Insomnia Relief (AIR) | Sleep Education (SE)
Started | 19 | 17
Completed | 17 | 16
Not Completed | 2 | 1
Not completed — Exclusion criterion met during the trial | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: 36 Veterans were randomized to treatment. 34 Veterans' data were retained for data analysis. Two Veterans' data were excluded because exclusion criteria were met during the trial.
Groups:
- Total: Total of all reporting groups
Arm/Group | Apnea and Insomnia Relief (AIR) | Sleep Education (SE) | Total
Number analyzed (Participants) | 18 | 16 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.06 (12.19) | 49.44 (12.16) | 50.29 (12.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 16 | 16 | 32
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: One participant did not specify their race/ethnicity.
  Participants
    Race/ethnicity: number analyzed (Participants) | 17 | 16 | 33
    Race/ethnicity: Caucasian/White | 11 | 8 | 19
    Race/ethnicity: Black or African American | 2 | 2 | 4
    Race/ethnicity: Asian | 2 | 3 | 5
    Race/ethnicity: Hispanic or Latino | 1 | 2 | 3
    Race/ethnicity: Other | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18 | 16 | 34

OUTCOME MEASURES:

1. Primary Outcome: World Health Organization Quality of Life (WHOQOL-BREF)
Description: This 26-item self-report questionnaire measures the following four broad domains: physical health, psychological health, social relationships, and environment. Each item has five response options, with higher scores indicating greater health. Mean scores are calculated for each domain and then multiplied by four (range of 4-20 for each domain) to enable comparisons with the WHOQOL-100. The primary outcome is the psychological domain.
Time Frame: Change from baseline to 1 week post-treatment (after 6 weeks)
Population: An intent-to-treat analysis was conducted using all available data from eligible participants who started treatment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Apnea and Insomnia Relief (AIR) | Sleep Education (SE)
Number analyzed (Participants) | 18 | 16
units on a scale
  Baseline | 11.26 (1.91) | 9.75 (2.95)
  Post-Treatment: number analyzed (Participants) | 17 | 15
  Post-Treatment | 12.78 (2.04) | 10.84 (2.80)

2. Primary Outcome: World Health Organization Quality of Life (WHOQOL-BREF)
Description: as for outcome 1
Time Frame: Change from baseline to 3 months after treatment ends
Population: An intent-to-treat analysis was conducted using all available data from eligible participants who started treatment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Apnea and Insomnia Relief (AIR) | Sleep Education (SE)
Number analyzed (Participants) | 18 | 16
units on a scale
  Baseline | 11.26 (1.91) | 9.75 (2.95)
  3-Month Follow-Up: number analyzed (Participants) | 17 | 14
  3-Month Follow-Up | 12.47 (2.55) | 10.71 (2.39)

3. Secondary Outcome: Functional Outcomes of Sleep Questionnaire (FOSQ-10)
Description: This 10-item self-report measure evaluates functional status. In particular, items prompt participants to rate the extent to which they experience difficulty completing various tasks due to sleepiness or fatigue. Responses to items range from 0 to 4. Total scores range from 5-20. Higher scores indicate better functioning.
Time Frame: Change from baseline to 1 week post-treatment (after 6 weeks)
Reporting Status: Not Posted

4. Secondary Outcome: Functional Outcomes of Sleep Questionnaire (FOSQ-10)
Description: as for outcome 3
Time Frame: Change from baseline to 3 months after treatment ends
Reporting Status: Not Posted

5. Secondary Outcome: Insomnia Severity Index (ISI)
Description: This seven-item self-report scale assesses severity of insomnia. Responses to items range from 0 to 4. Total scores range from 0 to 28. Higher scores indicate greater symptom severity.
Time Frame: Change from baseline to 1 week post-treatment (after 6 weeks)
Reporting Status: Not Posted

6. Secondary Outcome: Insomnia Severity Index (ISI)
Description: as for outcome 5
Time Frame: Change from baseline to 3 months after treatment ends
Reporting Status: Not Posted

7. Secondary Outcome: Total Sleep Time (Actigraphy-based)
Description: An actigraph will be used to determine total sleep time. An actigraph is a validated objective sleep measurement device commonly used outside the laboratory setting to detect movement and infer sleep and wake based on wrist activity.
Time Frame: Change from baseline to 1 week post-treatment (after 6 weeks)
Reporting Status: Not Posted

8. Secondary Outcome: CPAP Adherence
Description: Average daily CPAP use.
Time Frame: Past 7 days, at 1 week after treatment ends
Reporting Status: Not Posted

9. Secondary Outcome: CPAP Adherence
Description: Average daily CPAP use.
Time Frame: Past 7 days, at 3 months after treatment ends
Reporting Status: Not Posted

10. Secondary Outcome: Clinician Administered PTSD Scale for DSM-5 (CAPS-5)
Description: This 30-item semi-structured interview provides a dimensional and categorical measure of PTSD. The severity score is based on frequency and intensity of PTSD symptoms. Categorically, it determines presence of both lifetime and current PTSD. Current and lifetime PTSD will be assessed at pre-treatment. Only current PTSD will be assessed at post-treatment. This interview also assesses the onset and duration of symptoms, distress, impact of symptoms on functioning (social and occupational), change in symptoms since a previous administration, response validity, and dissociative subtype of PTSD.
Time Frame: Change from baseline to 1 week post-treatment (after 6 weeks)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 5 months
Arm/Group | Apnea and Insomnia Relief (AIR) | Sleep Education (SE)
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/16
Other Adverse Events (participants affected / at risk) | 0/18 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-10-22): https://cdn.clinicaltrials.gov/large-docs/96/NCT04007796/Prot_SAP_001.pdf
  • Informed Consent Form (2020-07-21): https://cdn.clinicaltrials.gov/large-docs/96/NCT04007796/ICF_000.pdf